CLINICAL TRIAL: NCT04805918
Title: An Ounce of Prevention is Worth a Pound of Cure: A Randomised Controlled Trial of Pedagogues Promoting Positive Parenting in a Home-visiting Program in At-risk Families
Brief Title: Pedagogues Promoting Positive Parenting in a Home-visiting Program in At-risk Families: A RCT of VIPP-SD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Væver, PhD Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Danish VIPP-SD RCT study
Record Dates: First submitted 2021-03-12; First posted 2021-03-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Behavior Problems in Early Childhood
Keywords: Selected early intervention; parental sensitivity and sensitive discipline; child externalizing behavior; pedagogues

STUDY DESIGN:
Intervention Model Description: The study population will be randomly allocated in the ratio 1:1 to either VIPP-SD or CAU. The randomization is stratified by municipality. A computer-generated list of random numbers is used for the allocation of participants. The allocation list is created using block randomization with block sizes of 10. The allocation sequence is generated by an investigator with no clinical involvement in the project.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor: The individual who evaluates the video-based outcome(s) of interest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIPP-SD (Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline). (Experimental): The VIPP-SD includes seven sessions of 1½-2 hours each with an 2-4 weeks interval VIPP-SD is delivered by a VIPP-SD trained pedagogue and takes place in the family home and the targeted parent and child are videotaped during daily interactions. The intervener studies the video and prepares feedback. During the sessions, the intervener and parent review the video together and the intervener provides their feedback according to the VIPP-SD protocol.
  Interventions: Behavioral: VIPP-SD
- Care as ususl (Active Comparator): The existing standard practices for parents of 2-6 year old children identified to be at risk for developing externalizing problems in the participating municipalities will be the active control condition. These vary in content and duration in the municipalities. Likewise, CAU may change during the project period. The exact content and duration of CAU interventions as well as participants' adherence to treatment will be described as precisely as possible.
  Interventions: Behavioral: VIPP-SD

INTERVENTIONS:
Behavioral: VIPP-SD — Parenting program

SUMMARY:
Supportive parenting is a strong predictor of positive outcomes for children, and harsh parenting is a risk factor for child development, especially for the child developing externalizing problems (overactive, oppositional, and aggressive behavior). Externalizing problems in preschoolers are predictive of a variety of problems in later childhood. Thus, parents are key targets for change in preventive programs with children at risk for developing externalizing problems. More than 95% of 2-6 year old Danish children spend an average of 7.5 hours, 5 days a week in a daycare setting, thus pedagogues are key frontline staff in the promotion of parental abilities and early childhood mental health. However, a recent Danish study shows that pedagogues experience a need for systematic skills and methods for intervening in families with a child at risk. Attachment-based programs enhancing parental sensitivity and parental sensitive discipline show promising results. This efficacy study examines the Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline (VIPP-SD)delivered by 22 VIPP-SD trained pedagogues at home-visits to 120 families with a child (1-6 years) identified to be at risk. Pedagogues are supervised by four VIPP municipality psychologists, thus promoting the cross-disciplinary collaboration. The results will point to future identification of families that may (and may not) profit from a pedagogue delivered VIPP-SD intervention, as well as to revise the intervention in order to maximizing its effect, i.e. point to changes to tailor intervention to the particular needs of different families in a Danish context.

ELIGIBILITY:
Inclusion Criteria:

* Child 2-6 year old
* Parent must be more than 18 years old
* Parent must speak and understand Danish
* Family must live in the municipalities of Frederiksberg or Roskilde - and having no intentions of moving out of the municipality before after the intervention has ended
* Parent can attend other treatment initiatives
* Child must attend a daycare center in one of the two municipalities
* Child must be at risk of developing externalizing behavior, i.e. showing signs of overactive, oppositional, and aggressive behavior.

Exclusion criteria

* Sexual or physical abuse by parent
* Parental drug or alcohol abuse
* Child diagnosis of autism
* Child is not considered at risk of developing externalizing behavior problems, but may have other problems, such as delayed language or motordevelopment etc

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Parental attitudes toward sensitivity and sensitive discipline (ATSSD) | Through study completion, an average of 6 months
  Questionnaire regarding parents' attitudes towards parenting (Bakermans-Kranenburg & Van IJzendoorn, 2003)

SECONDARY OUTCOMES:
Parenting Daily Hassles (PDH) | Through study completion, an average of 6 months
  Parenting Daily Hassles scale where parents are asked to rate 20 minor parenting stresses that often occur in families with small children (Crnic & Greenberg, 1990).
Parenting Stress | Through study completion, an average of 6 months
  via self-report using Parenting Stress IndexTM, Fourth Edition Short Form (PSI-4-SF;Abidin, 1995)
Parental Mentalizing | Through study completion, an average of 6 months
  self-report using the Parental Reflective Functioning Questionnaire (PRFQ; Luyten, Mayes, Nijssens, & Fonagy, 2017).
Family functioning | Through study completion, an average of 6 months
  self-report using the McMaster Family Assessment Device (FAD), the six item version (de Haan et al., 2015)
Parental symptoms of anxiety | Through study completion, an average of 6 months
  Anxiety symptoms will be assessed with GAD-7, which is a 7-item screening questionnaire for generalized anxiety disorder (Spitzer, Kroenke, Williams & Löwe, 2006).
Parental behavioral sensitivity and sensitive discipline | Through study completion, an average of 6 months
  Parental sensitivity will be coded from video recordings of parent-child free play. Coding will be conducted using Coding Interactive Behavior (CIB) (Feldman, 1998).
  Parental sensitive discipline will be coded from video recordings of a "don't touch task" and a "clean-up task". Coding procedure will be based on guidelines from Kuczynski et al., 1987 and Van der Mark et al., 2002.
Child behavior problems | Through study completion, an average of 6 months
  This is measured using the Strengths and Difficulties questionnaire (SDQ), which is completed by both parents and pedagogues (Goodman, 1997; Danish version by Niclasen et al., 2012).
Child socio-emotional development | Through study completion, an average of 6 months
  Child socio-emotional development is assessed via parental report using the Ages & Stages Questionnaires®: Social-Emotional, Second Edition (ASQ®:SE-2) (Squires, Bricker, & Twombly, 2015).
Parental symptoms of depression | Through study completion, an average of 6 months
  Depression symptoms will be assessed with PHQ-9, which is a 9-item questionnaire to monitor the severity of depression symptoms (Kroenke, Sptizer & Williams, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: mette væver, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Center for Early Interventions and Family Studies, Department of Psychology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No